CLINICAL TRIAL: NCT00256789
Title: Combination of Weekly Radiation and Docetaxel for Locally Advanced Non Small Cell Lung Cancer: A Feasibility Study
Brief Title: Once Weekly Radiation for Lung Cancer With Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Oncology Research Associates (Other)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hypo 1
Record Dates: First submitted 2005-11-18; First posted 2005-11-22 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2005-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC, Non-Small Cell Lung Cancer,Weekly Radiation, Taxotere
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiation; Drug Therapy

INTERVENTIONS:
Procedure: Radiation
Drug: Chemotherapy

SUMMARY:
This program is designed for the treatment of patients with advanced non-small cell lung cancer. The study is designed for patients whose cancer is too advanced and therefore cannot be operated with the goal of completely removing the cancer. Patients at this stage of their disease traditionally receive radiation therapy or chemotherapy or both treatments in succession. Recently, the administration of both methods of treatment has been employed and preliminary studies indicate somewhat better results. Specifically, a new class of chemotherapy agents called taxanes used in combination with radiation therapy appear promising as determined in small studies. However, the best treatment for this type of cancer has not been established yet. One goal of this study is to investigate if the combination of the new drug Taxotere (a drug belonging to the taxane class) given on the day of the radiation is well tolerated and will result in enhanced shrinkage of the cancer compared to traditional radiation therapy. In this study the radiation will be given on one day, rather than divided over five days per week (Monday through Friday) as in previous studies. Previous research has shown that both equal in how effective they are in treating lung cancer. The study will use the drug Taxotere in conjunction with radiation therapy. Taxotere is an approved medicine by the United States Food and Drug Administration for the treatment of lung cancer.

The purpose of this study is to evaluate if the chemotherapy drug Taxotere administered once weekly together with concurrent radiation on the same day is effective in shrinking non-small cell lung cancer. This trial will also investigate how well this treatment is tolerated and what effects this treatment will have on the everyday life and activities of participants.

DETAILED DESCRIPTION:
40 patients with locally advanced and metastatic NSCLC will be enrolled (stages III and IV) and treated once per week for a total of 12 cycles (12 weeks) according to the schedule outlined below.

Chemotherapy: The suggested phase II dose for weekly Taxotere with concomitant standard chest radiotherapy was determined to be 20mg/m2. In our unpublished phase I clinical trial, we found 35 mg/m2 to be well tolerated and therefore this dose is chosen for this phase II study. The drug will be administered intravenously on the same day as the radiation. All patients will be premedicated 12 hours prior to chemotherapy with Decadrone. Patients will be followed and evaluated weekly by a physician.

Radiation therapy: Although radiation was delivered differently in previous Taxotere based combined modality studies, the total radiation dose remains the same. Treatment will be given to a large field with a 2-3 cm tumor margin. All involved or suspicious nodal areas will be radiated as well. To reduce volume toxicity, the "field within a field" technique will be employed. Tumor and involved nodes will receive 200 cGy + 300 cGy. A total of 12 treatments will be administered in weekly, single sessions. Total treatment will be 6000 cGy. Radiation treatment will be administered 24 hours after Taxotere infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologic evidence of NSCLC.
2. Should the patient have a history of another malignancy or a second malignancy be present or discovered, subjects will only be eligible if the NSCLC is determined by the PI to be the more life-threatening disease and the other malignancy would not have otherwise a significant impact on the subjects life-expectancy (e.g. basal cell carcinoma of skin, remote history of early stage breast cancer surgically cured).
3. All patients must have surgically incurable disease, i.e. locally advanced disease (stage III A or III B) or metastatic stage IV.
4. Performance status of 0 to 2 (ECOG Criteria).
5. Patients should have an absolute granulocyte count > 1500/mm3 and a platelet count > 100,000/mm3.
6. Patients should have adequate hepatic function as indicated by a serum bilirubin < upper limit of normal (ULN); ALT and AST <2.5 ULN if alkaline phosphatase is < ULN. Alkaline phosphatase may be up to 4 x ULN if transaminases are < ULN. However, patients who have both transaminase elevation > 1.5 x ULN and alkaline phosphatase > 2.5 x ULN are not eligible for this study.
7. Patients should have at least a predicted FEV1 of 30%.
8. Patients with active ischemic heart disease (NYHA Class III or IV), congestive heart failure, symptomatic arrythmias, or a recent history of a myocardial infarction are excluded.
9. Patients with pre-existing neuropathy (> grade 1) are not eligible for this study.
10. No other serious concurrent medical illness or active infection which would jeopardize the ability of the patient to receive with reasonable safety the chemotherapy and surgery program outlined in this protocol is allowed.
11. Signed informed consent: each patient must be aware of the neoplastic nature of his/her disease and willingly consent to participate in the study after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side effects, risks, and discomforts.
12. Pregnant women and nursing mothers are ineligible. Women of child-bearing potential must have a negative pregnancy test. Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for three months thereafter.
13. Patients with a history of severe hypersensitivity reaction to TaxotereÒ or other drugs formulated with polysorbate 80 must be excluded.
14. Patients must be at least 18 years old.

    -

    Exclusion Criteria:

    Not falling into the eligibility criteria outlined above

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-09; Primary Completion 2003-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Feasibility

SECONDARY OUTCOMES:
Toxicity, Safety, Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Paul Schwarzenberger, MD, Principal Investigator — Mobile Infirmary Hospital, Mobile, AL
Locations (1):
- Cancer Center and Mobile Infirmary Hospital, Mobile, Alabama, United States

REFERENCES:
- [Background] Slawson RG, Salazar OM, Poussin-Rosillo H, Amin PP, Strohl R, Sewchand W. Once-a-week vs conventional daily radiation treatment for lung cancer: final report. Int J Radiat Oncol Biol Phys. 1988 Jul;15(1):61-8. doi: 10.1016/0360-3016(88)90347-1. PMID 2839442
- [Background] Salazar OM, Slawson RG, Poussin-Rosillo H, Amin PP, Sewchand W, Strohl RA. A prospective randomized trial comparing once-a-week vs daily radiation therapy for locally-advanced, non-metastatic, lung cancer: a preliminary report. Int J Radiat Oncol Biol Phys. 1986 May;12(5):779-87. doi: 10.1016/0360-3016(86)90036-2. PMID 3519551
- [Background] Salazar OM, Van Houtte P, Rubin P. Once-a-week radiation therapy for locally advanced lung cancer. Final report. Cancer. 1984 Aug 15;54(4):719-25. doi: 10.1002/1097-0142(1984)54:43.0.co;2-s. PMID 6744205